CLINICAL TRIAL: NCT06401837
Title: Circadian Based Acupressure Therapy on Post-stroke Fatigue, Depression, and Sleep Disturbances in Ischemic Stroke Patients Undergoing Rehabilitation
Brief Title: Acupressure Therapy on Post-stroke Fatigue, Depression, and Sleep Disturbances in Ischemic Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen-Chun Liao, Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH111-REC2-070
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Cytokine; Circadian Rhythm; Acupressure; Post-stroke Fatigue; Sleep; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure application ( AA ) group (Experimental): Patients in the AA group will have the circadian based acupressure application twice a day, 5 days per week for 2 weeks. Acupressure application will be performed in the morning after one hour of breakfast and in the evening 1-2 hour before bedtime by a nurse well-trained with Chinese medicine nursing during the first week.
  Interventions: Behavioral: Circadian based acupressure application
- Routine care control (RC) group (No Intervention): Patients in the RC group will get routine care as usual for rehabilitation. The ambient light at night will keep as dark or dim (<30 lux) as well. The same education program for circadian-based life style as the AA group will be provided to patients and caregivers too.

INTERVENTIONS:
Behavioral: Circadian based acupressure application — Acupoints include three points in hand: PC6 Neiguan, LI4 Hegu, HT7 Shenmen; two points in leg: SP6 Sanyinjiao & ST36 Zusanli; and one point in back: DU14 Dazhui will be selected. The nurse will also teach patients and their caregiver how to apply acupressure on these acupoints. Self-administered acupressure application on the above acupoints will be performed and followed in the second week. A rehabilitation program and routine care will be scheduled as usual except for acupressure.
  Arms: Acupressure application ( AA ) group

SUMMARY:
Post-stroke fatigue (PSF) was defined as 'a subjective feeling of physical and/or mental exhaustion that is unrelated to exertion and does not typically improve with rest'. About 25~85% of first stoke patients had PSF in the first year. Literature review from animal studies suggested the mechanism of post-stroke fatigue may be due to prolonged production of inflammatory cytokines process after stroke. Acupuncture therapy which regulates the inflammatory process may have the potential to ameliorate fatigue symptoms alone with sleep disturbance after stroke. Acupressure which stimulating the same acupoints by manually pressure may make it easy to perform in anytime and anywhere. The effect of circadian based acupressure application on post-stroke fatigue and sleep disturbances need be further examined. The purpose of this two-year study is to

(1) explore the distribution of inflammatory cytokines (blood and urine IL-1β, IL-6, TNF-α, IL-8) and post-stroke fatigue and sleep, and (2) examine the effect of circadian-based acupressure application on the inflammatory cytokines (urine and blood IL-1β, IL-6, TNF-α, IL-8), and post-stroke symptoms fatigue and sleep) in ischemic stroke patients with post-stroke fatigue during rehabilitation. Ischemic stroke patients (N=240) will be assessed from the rehabilitation wards.

Patients with fatigue (FAS>=24) at assessment (n=78) will be further randomly assigned to the circadian based acupressure application group (AA), or the routine care control group (RC) for 2 weeks. Data of inflammatory cytokines (of IL-1β, IL-6, TNF-α, IL-8), post-stroke fatigue (Fatigue assessment scale), and sleep (Pittsburg Sleep Quality Index and consumer tracker) will be collected. Descriptive statistics, t-test, repeated measure ANOVA, linear/logistic regression or appropriate nonparametric equivalent will be used to compare pre-post differences and to compare differences between groups. Study results will provide information about the mechanism and effect of acupressure application on inflammation and post-stroke fatigue and sleep disturbances in ischemic stroke patients.

DETAILED DESCRIPTION:
This is a two-year project. Two groups, randomized controlled experimental design, will be used to examine the effects of circadian-based acupressure application on inflammatory cytokines and post-stroke symptoms (fatigue and sleep) in ischemic stroke patients with fatigue (Figure 3). Ischemic stroke patients with fatigue (FAS >=24) during the first 6 months of rehabilitation, who were screened from the primary assessment, will be randomly assigned to two groups: the circadian-based acupressure application group (AA ) and the routine care control group (RC). Each patient will receive a 2-week intervention according to their group.

Acupressure application (AA) group Patients in the AA group will have the circadian-based acupressure application twice a day, 5 days per week for 2 weeks. Acupressure application will be performed in the morning after one hour of breakfast and in the evening 12 hours before bedtime by a nurse well-trained in Chinese medicine nursing during the first week. Acupoints include three points in hand: PC6, LI4 Hegu, HT7 Shenmen; two points in leg: SP6 Sanyinjiao & ST36 Zusanli; and one point in back: DU14 Dazhui will be selected. The nurse will also teach patients and their caregivers how to apply acupressure on these acupoints. Self-administered acupressure application on the above acupoints will be performed and followed in the second week. A rehabilitation program and routine care will be scheduled as usual except for acupressure. During nighttime, ambient light will remain dark or dim (<30 lux). Education programs for circadian-based lifestyle and acupressure applications will be provided to patients and caregivers.

Routine care control (RC) group: Patients in the RC group will get routine care as usual for rehabilitation. The ambient light at night will also keep as dark or dim (<30 lux). The same education program for a circadian-based lifestyle as the AA group will also be provided to patients and caregivers.

Outcomes of inflammatory cytokines, post-stroke fatigue, and sleep will be compared during(the 1st week) and after intervention (2nd week) between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 50 years old and above, both sex.
2. Diagnosed with stroke, ischemic.
3. Consciousness clear (GCS>=13)
4. Stable vital signs and neurological functional status with no or controlled complications (e.g., infection or gastrointestinal bleeding).
5. With fatigue (FAS >=24)

Exclusion Criteria:

1. Severe cognition impairment unable to give consent
2. Dysphasia
3. Ventilation use
4. Multiple diseases with unstable conditions
5. Receiving acupuncture therapy with the same acupoints.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokines | 10 cc of urine sample in the morning will be collected from each patient at baseline, and after 2 weeks of intervention.
  Cytokine concentrations of IL-1β, IL-6, IL-8 and TNF-a were measured in the plasma and urine using the human cytokine LINCO-plex multiplex bead array (Linco Research, St. Charles, MO, USA). The microspheres are incubated with standards, controls and samples in a 96-well microtiter filter plate for 1 h at room temperature. After washing with assay wash buffer, diluted biotinylated secondary antibody was added to the appropriate wells and incubated for 1 h. After washing, streptavidin-phycoerythrin was added to each well and incubated for 30 min. After a final wash, the plate was analyzed using the Luminex 100 analyzer (Luminex Corp., Austin, TX, USA) to determine the concentration of the cytokines.
Sleep | Patients wear a consumer tracker at baseline, 1st week during intervention, and after 2nd weeks of intervention for 24 hours each.
  Sleep pattern will be measured by a consumer tracker (Fitbit or Garmin). Patients will wear a tracker on their normal wrist for 24 hours continuously except taking showers. Analysis of sleep pattern will be performed including minute and percentage of total sleep time, awake time, light sleep, deep sleep, and REM sleep. Diary for waking behaviors such as exercise, watching TV, meals, drinks, and time for sun shine etc. and sleeping behaviors such as wake after sleep, will be collected to help analyze sleep patterns. Consumer tracker is show to have appropriate accuracy in measuring sleep (Haghayegh, Khoshnevis, Smolensky, Diller, & Castriotta, 2019) and mobility (Straiton et al., 2018).
Sleep quality | Patients will fill out the PSQI questionnaire at baseline, 1st week during intervention, and after 2nd weeks of intervention.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. The PSQI assessed habitual sleep of adults over a 1-month time interval with consists of nineteen self-rated questions that generates seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A global PSQI score is summed from each component to have a range of 0-21. Higher score indicates worse sleep quality. A post hoc cutoff score of 5 is the cut point to discriminate "good" or "poor" sleeper. The overall Cronbach's alpha values of the global PSQI for examining internal consistency reliability ranged from 0.77-0.83 (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989; Carpenter & Andrykowski, 1998; Doi et al., 2000). Sensitivity and specificity of the PSQI ranged from 80%-89.6% and 86.5%-86.6%, respectively (Buysse et al., 1989; Doi et al., 2000; Tsai et al., 2005).
Fatigue. | Patients will be measured at baseline, 1st weeks during intervention, and after 2nd weeks of intervention.
  Post-stroke fatigue will be measured by the Fatigue Assessment Scale (FAS) (Michielsen et al., 2003). It consists 10 self-rated descriptors regarding how patient feel with each item scored from one to five (1 = never, 2 = sometimes, 3= regularly, 4= often, 5= always). Items 4 and 10 require reversed scoring. The higher score is associated with higher fatigue with a total score of 10-50. A cut-off of FAS >/=24 gave a sensitivity of 0.84 and specificity of 0.67 in classifying post-stroke fatigue on the FAS (Cumming & Mead, 2017). Patients will be measured at baseline, 1st weeks during intervention, and after 2nd weeks of intervention.

SECONDARY OUTCOMES:
Depression | Participants will be assessed by the GDS-15 at baseline. Depression will serve as a covariate in this study.
  A Short Form Geriatric Depression Scale (GDS-15) will be used to assess patients' depression. The GDS-15 consists of 15 questions with 10 indicated the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicated depression when answered negatively. Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression. Participants will be assessed by the GDS-15 at baseline, and after 2nd weeks of intervention. Depression will serve as a covariate in this study.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hospital Taichung East Branch, Taichung
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No